CLINICAL TRIAL: NCT01576094
Title: Phase I Study of Two Inodilators in Neonates Undergoing Cardiovascular Surgery
Brief Title: Two Inodilators Postsurgery in Neonates
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz (Other)
Collaborators: Hospital Universitario La Paz (Other); Fondo de Investigacion Sanitaria (Other)
Responsible Party: Principal Investigator, Adelina Pellicer, Principal Investigator, Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MilevoNeo
Record Dates: First submitted 2012-03-31; First posted 2012-04-12 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Low Cardiac Output Syndrome
Keywords: congenital heart disease
MeSH Terms: conditions — Cardiac Output, Low; Heart Defects, Congenital | interventions — Milrinone; Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Milrinone (Active Comparator): Milrinone (MR) lactate 1 mg/ml: dose 1, starting immediately after central lines were placed and maintained for the duration of the surgical procedure; dose 2, on NICU admission; dose 3, after 2 hours of stability with dose 2, and maintained up to 48 hours. Accordingly, patients randomised to MR received 0.5 , 0.75 and 1 microg/kg per min
  Interventions: Drug: Milrinone
- Levosimendan (Active Comparator)
  Interventions: Drug: Levosimendan

INTERVENTIONS:
Drug: Milrinone — Before surgery, patients received milrinone (MR) (milrinone lactate 1 mg/ml). Intravenous continuous infusion of the study drug through a separate central line started intraoperatively and was increased step-wise at predefined time points: dose 1, starting immediately after central lines were placed and maintained for the duration of the surgical procedure; dose 2, on NICU admission providing the patient was in stable haemodynamic condition; dose 3, starting after 2 hours of stability with dose 2, and maintained up to 48 hours IND infusion started. Accordingly, patients randomised to MR received 0.5 , 0.75 and 1 microg/kg per min
  Other Names: cronotrope
  Arms: Milrinone
Drug: Levosimendan — Before surgery patients received levosimendan (levosimendan 2.5 mg/ml). Intravenous continuous infusion of the study drug through a separate central line started intraoperatively and was increased step-wise at predefined time points: dose 1, starting immediately after central lines were placed and maintained for the duration of the surgical procedure; dose 2, on NICU admission providing the patient was in stable haemodynamic condition; dose 3, starting after 2 hours of stability with dose 2, and maintained up to 48 hours IND infusion started. Accordingly, patients randomised to LEVO received 0.1 , 0.15 and 0.2 microg/kg per min, for doses 1, 2 and 3, respectively.
  Other Names: Simdax
  Arms: Levosimendan

SUMMARY:
Congenital heart defects are the most prevalent group of congenital malformations in newborns. Surgery-related low cardiac output syndrome (LCOS) could be one of the reason for the unfavourable outcome of this population. The early use of inodilators (INDs), specifically milrinone (MR), is proposed to reduce afterload and increase inotropism. Studies in the paediatric population appear to support a clinical usefulness of MR similar to that observed in adults. Levosimendan (LEVO) is a novel class IND developed for the treatment of heart failure. Experience with LEVO in paediatric patients is scarce. The purpose of this study was to systematically test the efficacy and safety of milrinone (MR) and levosimendan (LEVO) in newborns undergoing cardiovascular surgery with cardiopulmonary bypass (CPB). Given the uncertainty about LEVO pharmacokinetics in neonates, the study was designed as a pilot, phase I feasibility study.

DETAILED DESCRIPTION:
Surgical repair is the primary therapy for congenital heart defects in the newborn. The neonatal cardiovascular system is at particular risk to develop the surgery-related low cardiac output syndrome (LCOS), thus vasoactive agents are routinely used in the postoperative management. Systematic research on the efficacy of these drugs is scarce in the newborn. As LCOS pathophysiology joints impaired myocardial contractility and the peripheral effects of ischemia/reperfusion injury on the endothelium, early use of inodilators (IND) are strongly recommended to reduce afterload and improve contractility. This study aims to test the equivalence in dose-dependent hemodynamic effects of 2 IND, Milrinone and Levosimendan, used early without loading dose in the preoperative period to prevent LCOS. By means of non-invasive technology the investigators will assess cardiac function (serial structural and functional echocardiography), the cerebral and peripheral perfusion and oxygenation (continuous near-infrared monitoring), cerebral function (continuous amplitude integrated EEG monitoring), will rule out CNS acquired lesions (serial transfontanelar echo-Doppler studies), and will follow up different biochemical markers of myocardial stress and apoptosis. Pharmacokinetic studies will be also performed.

ELIGIBILITY:
Inclusion Criteria:

* Newborns undergoing cardiovascular surgery who were in stable pre-operative haemodynamic condition
* Parental consent given

Exclusion Criteria:

* Parental consent refused
* Inodilators contraindicated

Max Age: 40 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Perfusion-oxygenation | NIRS evaluation started immediately after surgery and was maintained during 24 h. At 48 h after surgery, a new NIRS evaluation during 4 hours. At 96 h post-surgery, during 4h.
  Changes in cerebral and thigh oxyhaemoglobin (O2Hb), deoxyhaemoglobin (HHb), total haemoglobin (THb) and tissue oxygenation index (TOI). The cerebral and peripheral intravascular oxygenation as c∆HbD was also assessed.

SECONDARY OUTCOMES:
Blood gases | preoperative (baseline) and then one determination every 6 hours until 24 h post-surgery. One determination at 48h post-surgery. One determination at 96 h post-surgery.
Blood pressure | preoperative (baseline) to post-operative day 6.
temperature | preoperative (baseline) to post-operative day 6.
  central (axilla) and peripheral (foot) temperature
arterial oxygen saturation | preoperative (baseline) to post-operative day 6.
cooximetry | preoperative (baseline) and then one determination every 6 hours until 24 h post-surgery. One determination at 48h post-surgery. One determination at 96 h post-surgery.
lactate | preoperative (baseline) and then one determination every 6 hours until 24 h post-surgery. One determination at 48h post-surgery. One determination at 96 h post-surgery.
glucose | preoperative (baseline) and then one determination every 6 hours until 24 h post-surgery. One determination at 48h post-surgery. One determination at 96 h post-surgery.
haemoglobin concentration | preoperative (baseline) and then one determination every 6 hours until 24 h post-surgery. One determination at 48h post-surgery. One determination at 96 h post-surgery.
Biochemical markers | baseline, at 24h after surgery and on day 6 post-surgery
  Serum creatinine, N-terminal pro-brain natriuretic peptide (NT-proBNP), troponine I (TnI) and proinflammatory and antinflammatory factors [interleukin (IL) beta 1, IL 6, IL 7, IL 8, IL 10, and tumor necrotic factor alpha
Inodilators concentration | Basal, two hours after dose 2; and at 24 and 48h from the start of the IND infusion in infants receiving IND dose 3. Beyond that period (open study), daily samples were obtained for LEVO up to day 7 postsurgery, and at 10 and 14 days.
  Milrinone and Levosimendan plasma concentration
inotrope score | preoperative (baseline) and then one evaluation every 6 hours until 24 h post-surgery. At 48h post-surgery. At 96 h post-surgery.
  calculated according to Wernovsky

CONTACTS AND LOCATIONS:
Overall Officials: Adelina Pellicer, PhD, Principal Investigator — Dept. of Neonatology, La Paz University Hospital, Madrid; Joan Riera, MBE, Study Chair — Bio-Engineer and Nanotechnology Dept., Polytechnic University of Madrid; Paloma López, MD, Study Chair — Dept. of Neonatology, La Paz University Hospital, Madrid; María Carmen Bravo, PhD, Study Chair — Dept. of Neonatology, La Paz University Hospital, Madrid; Rosario Madero, MD, Study Chair — Division of Biostatistics, La Paz University Hospital, Madrid; Jesús Pérez-Rodríguez, PhD, Study Chair — Dept. of Neonatology, La Paz University Hospital, Madrid; Carlos Labrandero, MD, Study Chair — Dept. Paediatric Cardiology, La Paz University Hospital, Madrid; José Quero, PhD, Study Chair — Dept. of Neonatology, La Paz University Hospital, Madrid; Antonio Buño, PhD, Study Chair — Clinical Pathology Service, La Paz University Hospital, Madrid; Luis Castro, MD, Study Chair — Dept. Paediatric Anaesthesiology, La Paz University Hospital, Madrid; Fernando Cabañas, PhD, Study Chair — Dept. of Neonatology, La Paz University Hospital, Madrid
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

REFERENCES:
- [Background] Bravo MC, Lopez P, Cabanas F, Perez-Rodriguez J, Perez-Fernandez E, Quero J, Pellicer A. Acute effects of levosimendan on cerebral and systemic perfusion and oxygenation in newborns: an observational study. Neonatology. 2011;99(3):217-23. doi: 10.1159/000314955. Epub 2010 Sep 25. PMID 20881438